CLINICAL TRIAL: NCT04179799
Title: Diaphragm Stimulation After Human Spinal Cord Injury: Effects on Respiratory Neural Drive and Function
Brief Title: Diaphragm Pacing in Individuals With Spinal Cord Injuries
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB201902285; 1OT2OD023854 (NIH)
Record Dates: First submitted 2019-11-01; First posted 2019-11-27 (Actual); Results first posted 2024-05-30 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Cervical Spinal Cord Injury
Keywords: SCI; diaphragm pacing; respiratory impairment; diaphragm stimulation
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cervical SCI: Participants with acute, traumatic cervical spinal cord injuries (C-SCIs), classified according to the American Spinal Injury Association (ASIA) Impairment Scale (AIS) as A-C (complete SCI (A); motor complete SCI (B); motor incomplete with minimal motor function (C)), affecting C1-C6 spinal cord segments, and who have been scheduled to undergo implantation of a diaphragm pacer, or who have recently received (in past 5-days) implantation of intramuscular diaphragm pacing electrodes due to severe respiratory impairments and dependence on mechanical ventilation.
  Interventions: Device: Diaphragm Pacing

INTERVENTIONS:
Device: Diaphragm Pacing — Intramuscular stimulation of the diaphragm, or diaphragm "pacing' is achieved by laparoscopic placement of stimulation wires into each hemidiaphragm. Phrenic motor points on the diaphragm are mapped to optimize electrode placement. The electrodes are threaded into the diaphragm muscle and wire leads are externalized and attached to a stimulation controller.

SUMMARY:
This project will evaluate the effects of intramuscular diaphragm stimulation (pacing) and test the hypothesis that diaphragm pacing enhances neuromuscular diaphragm activation and respiratory function in adults with cervical spinal cord injuries (C-SCIs). The investigators will test the hypothesis by recording activity of the diaphragm from intramuscular pacing electrodes and conduct respiratory assessments in adults with intramuscular diaphragm pacing electrodes following acute, traumatic C-SCIs.

DETAILED DESCRIPTION:
Respiratory dysfunction is a leading cause of death in individuals with spinal cord injuries (SCIs). Nearly one-quarter of all SCI cases involve injury to the upper spinal cord segments which impairs neural activation of the diaphragm muscle and compromises breathing. Although mechanical ventilation can be life-saving after cervical SCI (C-SCI), it also triggers rapid and profound diaphragm muscle atrophy, thereby complicating (or even preventing) ventilator weaning. Intramuscular diaphragm stimulation, or diaphragm pacing, was developed to replace long-term ventilator support and is now used acutely post C-SCI (<4 months following injury) to promote ventilator weaning. This study will assess the effects of diaphragm stimulation on respiratory neural drive and breathing function in individuals with acute, traumatic C-SCI. Recording from these surgically implanted electrodes allows comparisons of electromyogram (EMG) recordings, in association with respiratory assessments, before and after short periods of diaphragm pacing to isolate the unique contribution of diaphragm pacing on neuromuscular diaphragm activation.

ELIGIBILITY:
Inclusion Criteria:

* Acute, traumatic cervical spinal cord injuries (C-SCIs), classified according to the American Spinal Injury Association (ASIA) Impairment Scale (AIS) as A-C
* Scheduled to undergo implantation of a diaphragm pacer, or who have recently received (in past 5-days) implantation of intramuscular diaphragm pacing electrodes due to severe respiratory impairments and dependence on mechanical ventilation

Exclusion Criteria:

* Progressive neuromuscular diseases such as multiple sclerosis and myasthenia gravis
* History of neurologic injuries such as stroke or prior SCI
* Chest wall injuries or deformities likely to influence breathing
* Pregnancy
* Cognitive impairments limiting study participation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute, traumatic C-SCIs, scheduled to receive intramuscular diaphragm pacing OR who have recently received a diaphragm pacer (within past 5-days) will be recruited from UF Health Shands Jacksonville, a Level-1 trauma hospital serving North Florida.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2020-01-10 (Actual); Primary Completion 2022-08-20 (Actual); Study Completion 2022-08-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emily Fox, PT, PhD, Principal Investigator — University of Florida
Locations (1):
- UF Health - Jacksonville, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cervical SCI
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Cervical SCI
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 2
Age, Continuous [Mean (Full Range); unit: years] | 48 [35 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Change in Electromyogram (EMG)
Description: Neuromuscular activation of the diaphragm will be assessed by recording diaphragm EMGs from the surgically-implanted intramuscular stimulating electrodes. This approach will allow for comparisons of EMG recordings across time. EMGs will be recorded during non-stimulated respiration (diaphragm pacer turned off) and simultaneously with assessments of respiratory function.
Time Frame: Baseline up to 24 hours
Population: Data not obtained from 3 participants. Data recorded during quiet breathing from 3 of 6 participants, 24hrs after use of diaphragm pacing.
Measure: Mean (Standard Deviation); unit: mV
Arm/Group | Cervical SCI
Number analyzed (Participants) | 3
mV | -.0031 (.043)

2. Primary Outcome: Change in Maximal Inspiratory Pressure (MIP)
Description: The Maximum Inspiratory Pressure (MIP) is measured by a device that applies an inspiratory load which provides a resistance. The MIP will be measured in cmH20 and assesses diaphragm strength. MIP will be recorded will be recorded during non-stimulated respiration (diaphragm pacer turned off).
Time Frame: Baseline up to 24 hours
Population: 3 of the 6 participants were unable to complete this outcome measure.
Measure: Mean (Standard Deviation); unit: cmH2O
Arm/Group | Cervical SCI
Number analyzed (Participants) | 3
cmH2O | .27 (3.2)

3. Primary Outcome: Change in Tidal Volume
Description: The measurement of Tidal Volume is performed through a simple spirometry and is measured in liters. Tidal Volume will be recorded during non-stimulated respiration (diaphragm pacer turned off).
Time Frame: Baseline up to 24 hours
Population: data were not obtained from 1 participant
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Cervical SCI
Number analyzed (Participants) | 5
liters | .02 (.15)

ADVERSE EVENTS:
Time Frame: 1 week
Arm/Group | Cervical SCI
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-02-03): https://cdn.clinicaltrials.gov/large-docs/99/NCT04179799/Prot_SAP_000.pdf
  • Informed Consent Form (2021-10-20): https://cdn.clinicaltrials.gov/large-docs/99/NCT04179799/ICF_001.pdf